CLINICAL TRIAL: NCT06271200
Title: Effects of Intensive Lifestyle Interventions (ILI) on Weight Loss and Cardiometabolic Risks in Obese Adults With Metabolic Syndrome: A Randomized Clinical Trial
Brief Title: Strategic Lifestyle Intervention for Metabolic Syndrome (SLIM-MET)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); Taichung Armed Forces General Hospital (Other Government)
Responsible Party: Principal Investigator, Wayne Huey-Herng Sheu, Vice President and Distinguished Investigator, National Health Research Institutes, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MG-113-GP-03
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome
Keywords: Weight loss; Intermittent fasting; 10,000 steps; Mobile App; Continuous glucose monitoring (CGM); GLP-1 receptor agonist; SGLT-2 inhibitor
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This study is a randomized, parallel-group, observer-masked clinical trial. A total of 200 obese participants with MetS will be enrolled. Eligible subjects will be randomly assigned to the ILI group or ULI group with an allocation ratio of 2:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive lifestyle intervention (Experimental): Participants in the ILI group will receive an intensive lifestyle program including time-restricted eating and increased physical activity.
  Interventions: Other: Strategic lifestyle and drug interventions
- Control (Other): Participants in the ULI group will maintain their usual lifestyle without intervention during the first 24 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Strategic lifestyle and drug interventions — Participants in the Intensive Lifestyle Intervention (ILI) group will follow a program including:
  1. time-restricted eating with a 16:8 pattern (eating within an 8-hour window, fasting for 16 hours),
  2. walking over 10,000 steps daily, and
  3. a daily calorie reduction of 500 kcal (with macronutrient distribution: 40-55% carbohydrates, 15-20% protein, 20-30% fat).
  Participants in the Usual Lifestyle Intervention (ULI) group will maintain their habitual meal timing.
  After the initial 24-week lifestyle program, ILI participants will be randomized (1:1) to receive either a GLP-1 receptor agonist (Rybelsus) or an SGLT-2 inhibitor (Forxiga) for 26 weeks, while continuing their lifestyle regimen. This phase will assess the impact of medication-with or without prior lifestyle intervention-on weight loss and liver fat. All participants will then be followed for an additional 52 weeks to evaluate long-term weight maintenance.
  Arms: Intensive lifestyle intervention
Other: Control — Participants in the ULI group will maintain their usual lifestyle without intervention during the first 24 weeks.
  After the initial 24-week usual lifestyle intervention, participants in the ULI group will be randomly assigned in a 1:1 ratio to receive either Rybelsus (GLP-1 receptor agonist) or Forxiga (SGLT-2 inhibitor) for a duration of 26 weeks. This phase aims to assess the effects of these medications on weight reduction and liver fat content without prior intensive lifestyle intervention. All participants will be followed for an additional 52 weeks to evaluate the long-term sustainability of weight loss.
  Arms: Control

SUMMARY:
This study is a randomized, parallel-group, observer-masked clinical trial. A total of 200 obese participants with MetS will be enrolled. Eligible subjects will be randomly assigned to the ILI group or ULI group with an allocation ratio of 2:1. The ILI group will be instructed to eat in 8 hours while fasting in 16 hours on daily basis over 24 weeks. Furthermore, enhanced daily physical activities with walking more than 10,000 steps will be implemented. The enrolled participants will be instructed to follow a diet with reduction of daily intake of 500 kcals per day. ILI group will be asked to use the Health2Sync mobile app to track self-measured outcomes and daily diet control. The investigators objectively measure step counts for participants of ILI group during 24-week intervention period using a wearable device (Fitbit Inspire 2). Participants are asked to attach the pedometer on their waist belt, except while bathing and sleeping. The ULI group will be instructed to follow habitual meal timing. In addition, all participants of both groups will receive the health education. Anthropometric, sociodemographic data, biochemical variables, and metabolic variables will be measured at baseline and during follow-up visit. DEXA and MRI of abdomen will be measured at baseline and during following up visits. The proposed trial is designed to provide 85% statistical power to detect a significant difference in changes in the metabolic syndrome severity score after reduction > 5% body weight over 24 weeks.

After completion of the initial 24-week lifestyle intervention, which often has limited weight loss efficacy when used alone, a second-phase intervention will be conducted from week 26 to week 52. Participants in both the ILI and ULI groups will be randomly assigned in a 1:1 ratio to receive one of two evidence-based oral weight control medications: a GLP-1 receptor agonist (Rybelsus) or an SGLT-2 inhibitor (Forxiga), for a duration of 26 weeks. The ILI group will continue with the daily 8-hour time-restricted eating and 16-hour fasting regimen, along with walking more than 10,000 steps per day. This phase aims to evaluate the effects of these two medications on weight reduction and liver fat content, with or without prior 26-week intensive lifestyle intervention. After the 26-week medication intervention, all participants will be followed for an additional 52 weeks to assess the sustainability of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged from ≥ 20 years to 65 years
* BMI 27.0 to 45.0 kg/m2 with metabolic syndrome by IDF definition

Exclusion Criteria:

* History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis
* Diagnosis of type 1 or type 2 diabetes and regular taking oral or injection hypoglycemic therapy
* History of malignant tumors with active managements.
* History of medullary thyroid carcinoma or diagnosis of multiple endocrine neoplasia syndrome type 2 (MEN 2)
* Serious liver dysfunction or chronic kidney disease (aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2)
* History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months History of severe gastrointestinal diseases or gastrointestinal surgery in the past 6 months
* History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity without regular managements.
* History of hypersensitivity to semaglutide or any component of RYBELSUS®, or history of severe hypersensitivity reactions to Forxiga, such as anaphylaxis or angioedema.
* Taking medications affecting weight or energy intake/energy expenditure in the last 3 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician
* Currently participating in weight loss programs or weight change in the past 3 months (>5% current body weight)
* Women who are pregnant or plan to become pregnant
* Patients who cannot be followed for 3 years (due to a health situation or migration)
* Patients who are unwilling or unable to give informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the metabolic syndrome severity score (Z score) after reduction > 5% body weight from baseline to 24 weeks | 24 weeks
  Metabolic syndrome severity will be measured by using Z score derived from Taiwan Biobank and Metabolic syndrome severity score (MSSS): MSSS calculation will be performed with the online tool "METS Severity Calculator" at ttp://publichealth.hsc.wvu.edu/biostatistics/metabolic-syndrome-severity-calculator/mets-severity-calculator/. The equations for calculation of MSSS are based on the NHANES study in the USA with the following arguments: age, race, gender, waist circumference, triglycerides (TG), high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, systolic blood pressure (SBP) and blood glucose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Huey-Herng Sheu, MD, PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- Institute of Molecular and Genomic Medicine, National Health Resesarch Institutes, Zhunan, Miaoli County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isomaa B, Almgren P, Tuomi T, Forsen B, Lahti K, Nissen M, Taskinen MR, Groop L. Cardiovascular morbidity and mortality associated with the metabolic syndrome. Diabetes Care. 2001 Apr;24(4):683-9. doi: 10.2337/diacare.24.4.683. PMID 11315831
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Mottillo S, Filion KB, Genest J, Joseph L, Pilote L, Poirier P, Rinfret S, Schiffrin EL, Eisenberg MJ. The metabolic syndrome and cardiovascular risk a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Sep 28;56(14):1113-32. doi: 10.1016/j.jacc.2010.05.034. PMID 20863953
- [Background] Hanley AJ, Karter AJ, Williams K, Festa A, D'Agostino RB Jr, Wagenknecht LE, Haffner SM. Prediction of type 2 diabetes mellitus with alternative definitions of the metabolic syndrome: the Insulin Resistance Atherosclerosis Study. Circulation. 2005 Dec 13;112(24):3713-21. doi: 10.1161/CIRCULATIONAHA.105.559633. PMID 16344402
- [Background] Hsu CN, Hou CY, Hsu WH, Tain YL. Early-Life Origins of Metabolic Syndrome: Mechanisms and Preventive Aspects. Int J Mol Sci. 2021 Nov 2;22(21):11872. doi: 10.3390/ijms222111872. PMID 34769303
- [Background] Schulz LO, Bennett PH, Ravussin E, Kidd JR, Kidd KK, Esparza J, Valencia ME. Effects of traditional and western environments on prevalence of type 2 diabetes in Pima Indians in Mexico and the U.S. Diabetes Care. 2006 Aug;29(8):1866-71. doi: 10.2337/dc06-0138. PMID 16873794
- [Background] Gami AS, Witt BJ, Howard DE, Erwin PJ, Gami LA, Somers VK, Montori VM. Metabolic syndrome and risk of incident cardiovascular events and death: a systematic review and meta-analysis of longitudinal studies. J Am Coll Cardiol. 2007 Jan 30;49(4):403-14. doi: 10.1016/j.jacc.2006.09.032. Epub 2007 Jan 12. PMID 17258085
- [Background] Tsao YC, Li WC, Yeh WC, Ueng SW, Chiu SY, Chen JY. The Association between Metabolic Syndrome and Related Factors among the Community-Dwelling Indigenous Population in Taiwan. Int J Environ Res Public Health. 2020 Dec 2;17(23):8958. doi: 10.3390/ijerph17238958. PMID 33276457
- [Background] Kalan Farmanfarma K, Kaykhaei MA, Adineh HA, Mohammadi M, Dabiri S, Ansari-Moghaddam A. Prevalence of metabolic syndrome in Iran: A meta-analysis of 69 studies. Diabetes Metab Syndr. 2019 Jan-Feb;13(1):792-799. doi: 10.1016/j.dsx.2018.11.055. Epub 2018 Dec 5. PMID 30641809
- [Background] Han TS, Lean ME. A clinical perspective of obesity, metabolic syndrome and cardiovascular disease. JRSM Cardiovasc Dis. 2016 Feb 25;5:2048004016633371. doi: 10.1177/2048004016633371. eCollection 2016 Jan-Dec. PMID 26998259
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Ryan DH, Yockey SR. Weight Loss and Improvement in Comorbidity: Differences at 5%, 10%, 15%, and Over. Curr Obes Rep. 2017 Jun;6(2):187-194. doi: 10.1007/s13679-017-0262-y. PMID 28455679
- [Background] Das SK, Balasubramanian P, Weerasekara YK. Nutrition modulation of human aging: The calorie restriction paradigm. Mol Cell Endocrinol. 2017 Nov 5;455:148-157. doi: 10.1016/j.mce.2017.04.011. Epub 2017 Apr 12. PMID 28412520
- [Background] Laaksonen DE, Lakka HM, Salonen JT, Niskanen LK, Rauramaa R, Lakka TA. Low levels of leisure-time physical activity and cardiorespiratory fitness predict development of the metabolic syndrome. Diabetes Care. 2002 Sep;25(9):1612-8. doi: 10.2337/diacare.25.9.1612. PMID 12196436
- [Background] Laule C, Atasoy D. Hunger potentiated. Cell Metab. 2023 May 2;35(5):723-725. doi: 10.1016/j.cmet.2023.04.005. PMID 37137283
- [Background] Perez-Martinez P, Mikhailidis DP, Athyros VG, Bullo M, Couture P, Covas MI, de Koning L, Delgado-Lista J, Diaz-Lopez A, Drevon CA, Estruch R, Esposito K, Fito M, Garaulet M, Giugliano D, Garcia-Rios A, Katsiki N, Kolovou G, Lamarche B, Maiorino MI, Mena-Sanchez G, Munoz-Garach A, Nikolic D, Ordovas JM, Perez-Jimenez F, Rizzo M, Salas-Salvado J, Schroder H, Tinahones FJ, de la Torre R, van Ommen B, Wopereis S, Ros E, Lopez-Miranda J. Lifestyle recommendations for the prevention and management of metabolic syndrome: an international panel recommendation. Nutr Rev. 2017 May 1;75(5):307-326. doi: 10.1093/nutrit/nux014. PMID 28521334
- [Background] Heymsfield SB, Harp JB, Reitman ML, Beetsch JW, Schoeller DA, Erondu N, Pietrobelli A. Why do obese patients not lose more weight when treated with low-calorie diets? A mechanistic perspective. Am J Clin Nutr. 2007 Feb;85(2):346-54. doi: 10.1093/ajcn/85.2.346. PMID 17284728
- [Background] Chaix A, Manoogian ENC, Melkani GC, Panda S. Time-Restricted Eating to Prevent and Manage Chronic Metabolic Diseases. Annu Rev Nutr. 2019 Aug 21;39:291-315. doi: 10.1146/annurev-nutr-082018-124320. Epub 2019 Jun 10. PMID 31180809
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Gill S, Panda S. A Smartphone App Reveals Erratic Diurnal Eating Patterns in Humans that Can Be Modulated for Health Benefits. Cell Metab. 2015 Nov 3;22(5):789-98. doi: 10.1016/j.cmet.2015.09.005. Epub 2015 Sep 24. PMID 26411343
- [Background] Chow LS, Manoogian ENC, Alvear A, Fleischer JG, Thor H, Dietsche K, Wang Q, Hodges JS, Esch N, Malaeb S, Harindhanavudhi T, Nair KS, Panda S, Mashek DG. Time-Restricted Eating Effects on Body Composition and Metabolic Measures in Humans who are Overweight: A Feasibility Study. Obesity (Silver Spring). 2020 May;28(5):860-869. doi: 10.1002/oby.22756. Epub 2020 Apr 9. PMID 32270927
- [Background] Lowe DA, Wu N, Rohdin-Bibby L, Moore AH, Kelly N, Liu YE, Philip E, Vittinghoff E, Heymsfield SB, Olgin JE, Shepherd JA, Weiss EJ. Effects of Time-Restricted Eating on Weight Loss and Other Metabolic Parameters in Women and Men With Overweight and Obesity: The TREAT Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1491-1499. doi: 10.1001/jamainternmed.2020.4153. PMID 32986097
- [Background] Pan WH, Flegal KM, Chang HY, Yeh WT, Yeh CJ, Lee WC. Body mass index and obesity-related metabolic disorders in Taiwanese and US whites and blacks: implications for definitions of overweight and obesity for Asians. Am J Clin Nutr. 2004 Jan;79(1):31-9. doi: 10.1093/ajcn/79.1.31. PMID 14684394
- [Background] Gurka MJ, Lilly CL, Oliver MN, DeBoer MD. An examination of sex and racial/ethnic differences in the metabolic syndrome among adults: a confirmatory factor analysis and a resulting continuous severity score. Metabolism. 2014 Feb;63(2):218-25. doi: 10.1016/j.metabol.2013.10.006. Epub 2013 Oct 24. PMID 24290837